CLINICAL TRIAL: NCT02685423
Title: Optimized Visual Recovery in Adult Human Amblyopia Through Binocular Deprivation
Brief Title: Light-deprivation Utilized to Mitigate Amblyopia
Acronym: LUMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: State University of New York College of Optometry (Other)
Collaborators: University of Maryland, College Park (Other); Nova Southeastern University (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ben Backus, Associate Professor, State University of New York College of Optometry
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUMA_758485; R21EY025398 (NIH)
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Amblyopia
Keywords: Amblyopia; Lazy Eye; Anisometropia
MeSH Terms: conditions — Amblyopia; Anisometropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visual Deprivation - 10 days (Experimental): 10 days of visual deprivation followed by vision training
  Interventions: Behavioral: Binocular deprivation 10 days; Behavioral: Vision training
- Vision Training Only (Active Comparator): Vision training without visual deprivation
  Interventions: Behavioral: Vision training

INTERVENTIONS:
Behavioral: Binocular deprivation 10 days — Research participants will be asked to live 10 days in an experimentally-controlled dark environment.
  Other Names: Dark exposure 10 days; Visual deprivation 10 days; Darkness sequestration 10 days; Dark rearing 10 days
  Arms: Visual Deprivation - 10 days
Behavioral: Vision training — Subjects will play a video game on their VR headset for 24 minutes per day, followed by 20 minutes of binocular experience with a brightness-reducing filter over the non-amblyopic eye.
  Other Names: Visual therapy; Vision therapy; Visual learning; Perceptual learning

SUMMARY:
Amblyopia is an impairment in spatial vision caused by asymmetry in the quality of visual input across the two eyes during childhood. It is difficult to treat in adulthood because the visual system becomes less "plastic" (able to learn) with age. The purpose of this study is to determine whether five to ten days of visual deprivation--living in complete darkness--can enhance plasticity in the visual cortex and thereby facilitate the learning that is needed to recover visual function in amblyopic adults.

DETAILED DESCRIPTION:
An asymmetry in the visual input across the eyes early in postnatal life causes amblyopia, the most common basis of uni-ocular blindness in humans. If uncorrected, amblyopia results in the unaffected eye controlling the binocular visual cortex, while the ability of the affected eye to stimulate cortical neurons may weaken to the point of functional blindness. Previous attempts to recover vision in adult amblyopes have had limited success, and the investigators propose this is due in large part to the significant reduction of synaptic plasticity that occurs during cortical development. The investigators propose that optimal recovery from amblyopia in adulthood is a two stage process that requires 1) the reactivation of plasticity in the adult amblyopic cortex (permissive step) and 2) focused visual experience to stimulate perceptual learning (instructive step).

The Elizabeth Quinlan lab at the University of Maryland has recently shown that binocular visual deprivation in adulthood enhances synaptic plasticity in the adult cortex of experimental animals in as little as three days. In addition, binocular visual deprivation prior to repetitive visual experience stimulates the recovery of spatial acuity in an animal model of deep amblyopia. Here the investigators propose to translate this finding to the treatment of amblyopia in humans. The investigators propose to use binocular visual deprivation to promote synaptic plasticity in the amblyopic visual cortex, followed by visual perceptual learning through vision therapy homework, to stimulate the recovery of visual function. While visual perceptual learning has been previously shown to enhance visual function in amblyopic adults, the gains are slow and modest. The investigators predict that "pre-treatment" of the amblyopic visual system with binocular visual deprivation will enhance the magnitude and/or time course of learning-induced recovery from amblyopia.

Twenty-four adult amblyopes, age 18 or older, will be recruited for the study. The investigators will exclude amblyopes with strabismus history because the treatment has not been designed to improve binocular alignment (motor fusion). Thus, amblyopes will be form deprivation amblyopes, especially form deprivation due to anisometropia, with moderate (20/30 to 20/80) or severe (20/100 to 20/400) acuity in the affected eye. Screening will include an extensive application, telephone interview of two personal references, comprehensive visual examination, and in-person interview.

Participants will be fitted with new ophthalmics if indicated and followed for several weeks to allow their amblyopia to stabilize. Their visual function will be assessed behaviorally and also by direct measurement of neural activity using visually evoked potentials (VEPs). Participants will be assigned to one of three groups. One group will be sequestered for zero days, one for five continuous days, and one for ten continuous days. Participants in the five or ten day sequestration groups will undergo sequestration in groups of two, three, or four. After sequestration visual function will again be assessed, both behaviorally and with VEP. All participants will then undergo 8 weeks (3 weeks before, 5 weeks after) of vision treatment for amblyopia, based on video game play. Vision testing will occur regularly during this period and for 10 months thereafter. A third VEP scan will be done at the end of the 8 week treatment period.

If successful, this work would transform therapy for adult amblyopia, and focus attention on the importance of incorporating methods to enhance synaptic plasticity as an adjunct to treatment. In addition, the insight gained from this work could be extended to strabismus, eye movement control disorders, and the restoration of optimal neural function after damage from stroke or other traumatic brain injury. The proposed experiment will also pioneer the use of binocular visual deprivation in human amblyopes, and develop standards for implementation, participant sequestration and care.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older
* Moderate (20/30 to 20/80) to severe (20/100 to 20/400) amblyopia with a visual acuity of 20/25 or better in the fellow eye
* Must live in or be commutable to the New York Metropolitan area

Exclusion Criteria:

* individuals with study-relevant phobias, anxiety disorders or other mental health disorders will be excluded, as will people taking anti-depressant or anti-anxiety drugs
* Must pass all stages of application process:

  * Review of full application
  * Phone interview
  * Telephone interview of two personal references
  * On-site eligibility screening evaluation
  * On-site complete ophthalmic evaluation
  * Criminal background check
  * On-site personal interview
  * Psychological exam
  * Physical exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Backus Lab Stereoacuity Assessment | Twice during the two weeks before sequestration to establish baseline, and again after sequestration: twice weekly for 2 weeks, then weekly for 2 weeks, then 2 times during the next month, monthly for 4 months, and then once every two months for 6 months
  4-alternative forced choice task in a stereoscope in the Backus lab. Data will by analyzed for each participant separately and aggregated by mean of change over time.
Change from baseline in contrast sensitivity function of amblyopic eye, fellow eye, and both eyes together, using the Sentio (R) CSF measurement device | Twice during the two weeks before sequestration to establish baseline, and again after sequestration: twice weekly for 2 weeks, then weekly for 2 weeks, then 2 times during the next month, monthly for 4 months, and then once every two months for 6 months
  15-20 minute procedure to assess CSF in the amblyopic eye, fellow eye, and using both eyes together. Data will by analyzed for each participant separately and aggregated by mean of change over time.
Change from baseline in acuity as measured using M&S Technologies automated ETDRS acuity test | Three times during the 2 months before sequestration to establish baseline, and again after sequestration: once a week for 2 weeks, then once a month for 2 months, then once every 3 months until study completion (at approximately 1 year)
  5-10 minute procedure to assess logMAR acuity. Data will by analyzed for each participant separately and aggregated by mean of change over time.

SECONDARY OUTCOMES:
Binocular motor fusion assessment | 3 times during the 2 months before sequestration, 4 times during 12 months after sequestration
  vergence range measured with standard clinical assessment (binocular fixation of varied-distance target). Data will not be aggregated.

OTHER OUTCOMES:
Daily self-report of visual hallucinations | Daily during 5 or 10 days of darkness sequestration
  Participants will make daily auditory recording to document any hallucinations (or other remarkable phenomena related to their mental or physical state).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Backus, PhD, Principal Investigator — Grad Ctr for Vision Research, SUNY College of Optometry
Locations (1):
- SUNY College of Optometry - Clinical Vision Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided